CLINICAL TRIAL: NCT01813188
Title: Phase II Clinical Trial of Tissue Engineering Based on the Use of Mononuclear Cells From Autologous Bone Marrow Seeded on Porous Tricalcium Phosphate Biomaterial in Patients With Pseudoarthrosis
Brief Title: Clinical Trial Based on the Use of Mononuclear Cells From Autologous Bone Marrow in Patients With Pseudoarthrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: Carlos III Health Institute (Other Government); Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCBO-PS
Record Dates: First submitted 2011-06-22; First posted 2013-03-18 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2014-03

CONDITIONS: Pseudoarthrosis
Keywords: Fractures; Bone; Stem Cells
MeSH Terms: conditions — Pseudarthrosis; Fractures, Bone | interventions — Dopamine beta-Hydroxylase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABM seeded onto a porous TCP and DBM (Experimental): ABM seeded onto a porous TCP and DBM
  Interventions: Procedure: ABM seeded onto a porous TCP and DBM
- autologous bone graft (Active Comparator): autologous bone graft
  Interventions: Procedure: autologous bone graft

INTERVENTIONS:
Procedure: ABM seeded onto a porous TCP and DBM — cells collection under sedation . 114 mL are obtained and processed through a ficoll gradient.
  Autologous bone marrow (ABM) cells seeded onto a porous tricalcium phosphate ceramic (TCP) and demineralized bone matrix (DBM)
  Arms: ABM seeded onto a porous TCP and DBM
Procedure: autologous bone graft — autologous bone graft
  Arms: autologous bone graft

SUMMARY:
The purpose of this clinical trial is to check the non-inferiority and lower morbidity of the use of bone marrow mononuclear cells seeded onto a porous matrix of calcium phosphate, for the consolidation of tibial bone defects (pseudoarthrosis), compared with autologous bone graft.

DETAILED DESCRIPTION:
An estimated 10% of closed fractures and between 35-45% in cases of open fractures, are at risk of developing a delay in the process of consolidation or a complete failure of it (pseudoarthrosis) depending on location , severity of trauma on bone, soft tissue and vascular structures Some of these cases are refractory to all treatment methods available today, requiring numerous interventions with the potential risk for recurrent infections that they carry. For this reason, its treatment remains a challenge for the orthopedic surgeon.

Recent advances in knowledge of cellular and molecular biology related to the mechanism of bone repair and biomaterials science have been joined in a new discipline called tissue engineering, its implementation in clinical practice is being done so progressive.

Cell therapy based on the use of adult stem cells (MSCs) derived from autologous bone marrow, introduces new applications for the repair of fractures including pseudoarthrosis and avascular bone necrosis.

Its mechanism of action does not focus only on their local action, but also in the release of signaling molecules with autocrine and paracrine action through recruitment and activation of endogenous MSCs to osteoblastic differentiation and bone tissue regeneration.

On the other hand, the seeding of MSCs on biomaterials (natural or synthetic) is more effective, to facilitate adherence, proliferation and extracellular matrix production in the area where implanted.

Today, the investigators can say that there are experimental and clinical evidence supporting the effectiveness of the method.

The investigators have designed a phase II clinical trial to check the feasibility of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Pseudarthrosis of tibia established any cause with at least 9 months.
* The pseudarthrosis is not to show signs of healing in the last 3 months.
* The pseudarthrosis subsidiary should not be solely osteosynthesis treatment.
* Age between 18 and 75 years.
* Serology Human Immunodeficiency virus (HIV), hepatitis B virus (HBV) and hepatitis C virus (HCV) negative.
* Negative pregnancy test in women of childbearing age.
* Patient sufficient guarantees of adherence to protocol.
* Signature written informed consent before a witness

Exclusion Criteria:

* Systemic infection.
* Septic pseudoarthrosis.
* Insufficient skin coverage at the site of nonunion.
* Vascular insufficiency in the affected limb.
* Pathological fracture.
* Concomitant psychiatric or neurological disease.
* Concurrent or prior malignancy treated with chemotherapy over a period of less than 1 year.
* Concomitant severe disease not well controlled.
* Inclusion in other clinical trials.
* Inability to understand the informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Time needed to repair the focus of necrosis measured by pain radiography | Baseline and every 14 days up to 180 days

SECONDARY OUTCOMES:
Pain scale | Baseline and every 14 days up to 180 days
Technical success | 6 months
  Understood as having been able to perform the implant of calcium phosphate matrix loaded with more than 100 million mononuclear cells
Morbidity | 6 months
  Infection of extraction points Pathological fracture of the extraction area Muscle hernia Stress fracture Infection of focus repaired Rupture of the focus fixture repaired Appearance of secondary malignancies
Absence of adverse events | 6 months
physical exploratory | Baseline and every 14 days up to 180 days
Analgesia Scale | Baseline and every 14 days up to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Luis Meseguer Olmo, MD,PhD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital UniversitarioVirgen de la Arrixaca, El Palmar, Murcia, Spain